CLINICAL TRIAL: NCT01723085
Title: Anti-Mullerian Hormone Levels Variations Following an Open Myomectomy
Brief Title: Anti-Mullerian Hormone Levels Before and After an Open Myomectomy
Status: Terminated | Type: Observational
Why Stopped: It has been put on hold for the moment due to logistic problems
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: AMH
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Anti-Mullerian Hormone
Keywords: Anti-Mullerian hormone; Myomectomy; Laparotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples collected to measure Anti-Mullerian hormone levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Open myomectomy: All patients belong to the same group Description includes the surgical technique

SUMMARY:
Anti-Mullerian hormone (AMH) is a marker for ovarian reserve. It is well known that ovarian surgery for endometriosis lowers Anti-Mullerian hormone, but little is known for other surgeries. We seek to investigate the hormone variations before and after an open myomectomy.

Hypothesis: Anti-Mullerian hormone levels drop following surgery but return to normal levels in a few months

ELIGIBILITY:
Inclusion Criteria:

* 18 to 42 years old
* Requiring open myomectomy for any indication

Exclusion Criteria:

* Incapable of informed consent
* Use of hormonal contraception or Gonadotropin-releasing hormone agonists in the past 3 months
* Woman over 42 years old
* Post-menopause women
* Positive B-human chorionic gonadotropin the day of surgery
* Ovarian surgery (at the same time)
* Pre-operative AMH below 0.3 ng/mL

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women 18 to 42 tears old Indication for myomectomy by laparotomy
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Anti-Mullerian Hormone levels variation | 6 months
  Anti-Mullerian Hormone levels before and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eric Himaya, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Hopital Saint-Luc, Montreal, Quebec, Canada